CLINICAL TRIAL: NCT01894919
Title: A Phase IIIb, Open Label, Multi Center Extension Study of V72_28 to Assess Antibody Persistence, and the Safety and Tolerability of a Booster Dose After the Completion of the Vaccination Course in Study V72_28
Brief Title: Antibody Persistence, and Safety and Tolerability of a Booster Dose of the Meningococcal B Vaccine After the Completion of the Vaccination Course in Study V72_28
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72_28E1; 2012-000657-30 (EudraCT Number)
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2018-05

CONDITIONS: Meningoccocal Disease; Meningococcal Meningitis
Keywords: Meningococcal B disease,; Antibody persistence
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (13):
- 2H3H511_V (Experimental): In the parent study V72_28 (NCT01339923), subjects received three primary doses and one booster dose of Bexsero® vaccine at 2.5, 3.5 and 5 months and at 11 months of age, respectively. The subjects in this group received a 5th dose of Bexsero® vaccine in the present study.
  Interventions: Biological: Bexsero® vaccine (1 dose at study month zero)
- 2H3H511_NV (No Intervention): In the parent study V72_28 (NCT01339923), subjects received three primary doses and one booster dose of Bexsero® vaccine at 2.5, 3.5 and 5 months and at 11 months of age, respectively. These subjects were evaluated only for persistence.
- 3H5_11_V (Experimental): In the parent study V72_28 (NCT01339923), subjects received two primary doses and one booster dose of Bexsero® vaccine at 3.5 and 5 months and at 11 months of age, respectively. These subjects received a 4th dose of Bexsero® vaccine in the present study.
  Interventions: Biological: Bexsero® vaccine (1 dose at study month zero)
- 3H5_11_NV (No Intervention): In the parent study V72_28 (NCT01339923), subjects received two primary doses and one booster dose of Bexsero® vaccine at 3.5 and 5 months and at 11 months of age, respectively. These subjects were evaluated only for persistence.
- 68_11_V (Experimental): In the parent study V72_28 (NCT01339923), subjects received two primary doses and one booster dose of Bexsero® vaccine at 6 and 8 months and at 11 months of age, respectively. These subjects received a 4th dose of Bexsero® vaccine in the present study.
  Interventions: Biological: Bexsero® vaccine (1 dose at study month zero)
- 68_11_NV (No Intervention): In the parent study V72_28 (NCT01339923), subjects received two primary doses and one booster dose of Bexsero® vaccine at 6 and 8 months and at 11 months of age, respectively. These subjects were evaluated only for persistence.
- 02_2_5_V (Experimental): In the parent study V72_28 (NCT01339923), these subjects received two catch-up doses of Bexsero® vaccine, two months apart. These subjects received a 3rd dose of Bexsero® vaccine in the present study.
  Interventions: Biological: Bexsero® vaccine (1 dose at study month zero)
- 02_2_5_NV (No Intervention): In the parent study V72_28 (NCT01339923), these subjects received two catch-up doses of Bexsero® vaccine, two months apart. These subjects were evaluated only for persistence.
- 02_6_10_V (Experimental): In the parent study V72_28 (NCT01339923), these subjects received two catch-up doses of Bexsero® vaccine, two months apart. These subjects received a 3rd dose of Bexsero® vaccine in the present study.
  Interventions: Biological: Bexsero® vaccine (1 dose at study month zero)
- 02_6_10_NV (No Intervention): In the parent study V72_28 (NCT01339923), these subjects received two catch-up doses of Bexsero® vaccine, two months apart. These subjects were evaluated only for persistence.
- NAIVE 123 (Experimental): Newly recruited naïve subjects who received two catch-up doses of Bexsero® vaccine, one month apart, in the present study.
  Interventions: Biological: Bexsero® vaccine (2 doses 1 month apart)
- NAIVE_4A (Experimental): Newly recruited naïve subjects who received two catch-up doses of Bexsero® vaccine, one month apart, in the present study.
  Interventions: Biological: Bexsero® vaccine (2 doses 1 month apart)
- NAIVE_4B (Experimental): Newly recruited naïve subjects who received two catch-up doses of Bexsero® vaccine, one month apart, in the present study.
  Interventions: Biological: Bexsero® vaccine (2 doses 1 month apart)

INTERVENTIONS:
Biological: Bexsero® vaccine (1 dose at study month zero)
  Arms: 02_2_5_V; 02_6_10_V; 2H3H511_V; 3H5_11_V; 68_11_V
Biological: Bexsero® vaccine (2 doses 1 month apart)
  Arms: NAIVE 123; NAIVE_4A; NAIVE_4B

SUMMARY:
The aim of this extension study is to explore the antibody persistence 24 to 36 months after the last dose of vaccine, in infants that received a two or three dose primary series plus a booster dose at 11 months of age, of the Novartis meningococcal B vaccine (Bexsero®) in groups I to III of the parent V72_28 study.

This study will also explore the antibody persistence 24 to 36 months after two catch-up doses of the Novartis meningococcal B vaccine (Bexsero®) administered in children (2 to 10 years old) in group IV of the parent V72_28 study.

ELIGIBILITY:
Inclusion Criteria:

For naïve subjects newly enrolled:

1. Healthy infants and children according to the following age groups:

   1. Healthy subjects from 35 to 47 months of age, (only applicable to group K) (The age window is defined as the first day the subject turns 35 months of age up to the day before the subject turns 48 months of age),
   2. Healthy subjects 4 to 7 years of age (only applicable to group L) (The age window is defined as the first day the subject turns 4 years of age up to the day before the subject turns 8 years of age).
   3. Healthy subjects 8 to 12 years of age (only applicable to group M) (The age window is defined as the first day the subject turns 8 years of age up to the day before the subject turns 13 years of age).
2. for whom a parent/legal guardian has given written informed consent after the nature of the study has been explained;
3. for whom a parent/legal guardian confirmed availability for the visit scheduled in the study;
4. in good health as determined by medical history, physical examination, clinical judgment of the investigator.

For Subjects who participated in the V72_28 study (Follow-on Subjects):

1. for whom a parent/legal guardian has given written informed consent after the nature of the study has been explained;
2. for whom a parent/legal guardian confirmed availability for the visit scheduled in the study;
3. in good health as determined by medical history, physical examination, clinical judgment of the investigator
4. who have completed the vaccination course in the V72_28 study and have received their last vaccination 24 to 36 months before enrollment in V72_28E1

Exclusion Criteria:

For naïve subjects newly enrolled:

1. History of any serogroup B meningococcal vaccine administration;
2. Previous known or suspected disease caused by N. meningitidis;
3. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection or colonization;
4. History of severe allergic reaction after previous vaccinations or hypersensitivity to any component of the vaccine;
5. Pregnancy or nursing (breastfeeding) mothers;
6. Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study. Oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide), intrauterine device, surgical sterilization, transdermal delivery, congenital sterility or sexual abstinence are considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods at least two months prior to study entry;
7. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from (for example):

   * Receipt of any chronic immunosuppressive therapy
   * Receipt of any chronic immunostimulants
   * Immune deficiency disorder, or known HIV infection
8. History of seizure, any progressive neurological disease or Guillain Barré Syndrome (exception: one self-limited febrile seizure is acceptable).
9. Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
10. Subject's parent(s) or legal guardian(s) are not able to comprehend and to follow all required study procedures for the whole period of the study.
11. Intent to participate in another clinical study during this study.
12. Family members and household members of study staff;
13. History or any illness/condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or pose additional risk to the subjects due to participation in the study.
14. Any significant chronic infection.
15. Any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).

For Subjects who participated in the V72_28 study (Follow-on Subjects):

Exclusion criteria are the same as for naïve subjects, with the exception of criterion 1.

Ages: 35 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 851 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (17):
- Hungary (9):
  - Site 34, General Pediatric Practice Somorjai, Debrecen, Bajcsi Ut 32
  - Site 35, Praxis Dr Eva Kovacs, Szeged, Csongradi Sgt 63
  - Site 36, General Practice Dr Edit Oszlacs, Szeged, Debreceni Utca 10-14
  - Site 37, Praxis Dr Julianna Kovacs, Bordány, Honved Utca 2
  - Site 31, General Practice Dr Olga Fekete, Miskolc, Kando Kalman Utca 1
  - Site 40, General Pediatric Practice Hacsek, Budapest, Poth Iren U 80
  - Site 30, General Practice Dr Simko, Miskolc, Selyemret U. 1.
  - Site 33, General Pediatric Practice Ujhelyi, Nyíregyháza, Szent Istvan U 10
  - Site 42, Praxis Dr Eszter Bari, Csongrád, Szentharomsag Ter 10
- Spain (8):
  - Site 15, Almería
  - Site 16, Almería
  - Site 20, Barcelona
  - Site 17, Madrid
  - Site 18, Madrid
  - Site 13, Pontevedra
  - Site 10, Santiago de Compostela
  - Site 14, Seville

REFERENCES:
- [Derived] Martinon-Torres F, Carmona Martinez A, Simko R, Infante Marquez P, Arimany JL, Gimenez-Sanchez F, Couceiro Gianzo JA, Kovacs E, Rojo P, Wang H, Bhusal C, Toneatto D. Antibody persistence and booster responses 24-36 months after different 4CMenB vaccination schedules in infants and children: A randomised trial. J Infect. 2018 Mar;76(3):258-269. doi: 10.1016/j.jinf.2017.12.005. Epub 2017 Dec 15. PMID 29253560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 study sites in Hungary and 8 study sites in Spain.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- 02_6_10_NV: In the parent study V72_28 (NCT01339923), these subjects received two catchup doses of Bexsero® vaccine, two months apart. These subjects were evaluated only for persistence.
Period: Overall Study
Arm/Group | 2H3H511_V | 2H3H511_NV | 3H5_11_V | 3H5_11_NV | 68_11_V | 68_11_NV | 02_2_5_V | 02_2_5_NV | 02_6_10_V | 02_6_10_NV | NAIVE 123 | NAIVE_4A | NAIVE_4B
Started | 98 | 47 | 89 | 43 | 81 | 39 | 32 | 36 | 91 | 90 | 100 | 55 | 50
Completed | 96 | 47 | 89 | 43 | 78 | 39 | 32 | 36 | 91 | 89 | 98 | 55 | 50
Not Completed | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other-Unspecified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2H3H511_V | 2H3H511_NV | 3H5_11_V | 3H5_11_NV | 68_11_V | 68_11_NV | 02_2_5_V | 02_2_5_NV | 02_6_10_V | 02_6_10_NV | NAIVE 123 | NAIVE_4A | NAIVE_4B | Total
Number analyzed (Participants) | 98 | 47 | 89 | 43 | 81 | 39 | 32 | 36 | 91 | 90 | 100 | 55 | 50 | 851
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.1 (0.2) | 3 (0.18) | 3.1 (0.23) | 3.1 (0.22) | 3.2 (0.29) | 3.2 (0.26) | 6.5 (1.15) | 6.7 (1.16) | 10.4 (1.43) | 10.4 (1.44) | 3.4 (0.29) | 5.8 (1.12) | 9.7 (1.38) | 5.6 (3.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 27 | 48 | 22 | 35 | 23 | 19 | 15 | 44 | 46 | 46 | 26 | 27 | 422
  Male | 54 | 20 | 41 | 21 | 46 | 16 | 13 | 21 | 47 | 44 | 54 | 29 | 23 | 429

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Activity Titers (hSBA) ≥ 4 or ≥ 5 Against Neisseria Meningitidis (N. Meningitidis) Serogroup B Strains
Description: The antibody persistence in subjects, 24 to 36 months after completion of Bexsero® vaccination course in the parent study according to different schedules, is presented in terms of the percentage of subjects in each vaccine group, with hSBA titers ≥ 4 for what concerns the H44/76, 5/99 and NZ98/254 strains, and hSBA titers ≥ 5 for M10713 strain, alongside with the corresponding antibody responses in age-matched vaccine naïve subjects at baseline.
  The functional bactericidal antibodies directed against serogroup B meningococcal were assessed by the Serum Bactericidal Assay (SBA) using human serum as the source of exogenous complement (hSBA).
Time Frame: 24-36 months after booster dose in the parent study; baseline for vaccine-naïve subjects
Population: Analysis was done on Full Analysis Set (FAS)-persistence: All subjects in the Enrolled Set who provide an evaluable serum sample at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- 2H3H511: Combined group 4D_2-11M/B + group 4D_2-11M - Subjects who received three primary doses and one booster dose of Bexsero® vaccine at 2.5, 3.5 and 5 months and at 11 months of age, respectively, in the parent study V72_28 (NCT01339923).
- 3H5_11: Combined group 3D_3-11M/B + group 3D_3-11M - Subjects who received two primary doses and one booster dose of Bexsero® vaccine at 3.5 and 5 months and at 11 months of age, respectively, in the parent study V72_28 (NCT01339923).
- 68_11: Combined group 3D_6-11Y/B + group 3D_6-11M - Subjects who received two primary doses and one booster dose of Bexsero® vaccine at 6 and 8 months and at 11 months of age, respectively, in the parent study V72_28 (NCT01339923).
- 02_2_5: Combined group 2D_2-5Y/B + group 2D_2-5Y- Subjects who received two catch-up doses of Bexsero® vaccine two months apart, at 2 and 5 years of age, respectively, in the parent study V72_28 (NCT01339923).
- 02_6_10: Combined group 2D_6-10Y/B + group 2D_6-10Y- Subjects who received two catch-up doses of Bexsero® vaccine two months apart, at 6 and 10 years of age, respectively, in the parent study V72_28 (NCT01339923).
Arm/Group | 2H3H511 | 3H5_11 | 68_11 | NAIVE 123 | 02_2_5 | NAIVE_4A | 02_6_10 | NAIVE_4B
Number analyzed (Participants) | 140 | 131 | 119 | 100 | 68 | 55 | 179 | 50
Percentage of subjects
  H44/76: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 178 | 50
  H44/76 | 51 [42.8 to 60] | 53 [43.8 to 61.5] | 61 [52 to 70.1] | 38 [28.5 to 48.3] | 52 [39.7 to 64.6] | 27 [16.1 to 41] | 58 [50.3 to 65.2] | 20 [10 to 33.7]
  5/99: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  5/99 | 84 [77.2 to 89.9] | 88 [80.9 to 92.9] | 93 [87.2 to 97.1] | 3 [0.6 to 8.5] | 79 [67.4 to 88.1] | 4 [0.44 to 12.5] | 85 [79.4 to 90.3] | 8 [2.2 to 19.2]
  NZ98/254: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  NZ98/254 | 45 [36.6 to 53.6] | 38 [29.8 to 47.1] | 56 [46.9 to 65.4] | 2 [0.24 to 7] | 29 [19 to 41.7] | 7 [2 to 17.6] | 50 [42.2 to 57.3] | 6 [1.3 to 16.5]
  M10713: number analyzed (Participants) | 127 | 111 | 109 | 93 | 65 | 53 | 173 | 49
  M10713 | 31 [22.8 to 39.5] | 36 [27.1 to 45.7] | 39 [29.4 to 48.3] | 37 [26.8 to 47.2] | 34 [22.6 to 46.6] | 38 [24.8 to 52.1] | 61 [53.0 to 68.0] | 55 [40.2 to 69.3]

2. Primary Outcome: Percentage of Subjects With hSBA Titers ≥ 8 Against N.Meningitidis Serogroup B Strains
Description: The antibody persistence in subjects, 24 to 36 months after completion of Bexsero® vaccination course in the parent study according to different schedules is presented in terms of the percentage of subjects in each vaccine group with hSBA titers ≥ 8, alongside with the corresponding antibody responses in age matched vaccine naïve subjects at baseline.
Time Frame: At 24-36 months after booster dose in the parent study: baseline for vaccine-naïve subjects
Population: Analysis was done on FAS-persistence: All subjects in the Enrolled Set who provide an evaluable serum sample at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2H3H511 | 3H5_11 | 68_11 | NAIVE 123 | 02_2_5 | NAIVE_4A | 02_6_10 | NAIVE_4B
Number analyzed (Participants) | 140 | 131 | 119 | 100 | 68 | 55 | 179 | 50
Percentage of subjects
  H44/76: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 178 | 50
  H44/76 | 28 [20.6 to 36.1] | 26 [18.7 to 34.3] | 32 [23.7 to 41.1] | 18 [11 to 26.9] | 24 [14.3 to 35.9] | 16 [7.8 to 28.8] | 34 [26.8 to 41.2] | 10 [3.3 to 21.8]
  5/99: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  5/99 | 80 [72.4 to 86.3] | 82 [74.8 to 88.5] | 89 [82 to 94.1] | 2 [0.24 to 7] | 73 [60.9 to 83.2] | 4 [0.44 to 12.5] | 66 [59.1 to 73.3] | 6 [1.3 to 16.5]
  NZ98/254: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  NZ98/254 | 21 [14.9 to 29.2] | 18 [12.1 to 26] | 29 [20.7 to 37.6] | 0 [0 to 3.6] | 15 [7.3 to 25.4] | 2 [0.05 to 9.7] | 28 [21.5 to 35.1] | 0 [0 to 7.1]
  M10713: number analyzed (Participants) | 127 | 111 | 109 | 93 | 65 | 53 | 173 | 49
  M10713 | 24 [16.5 to 32] | 22 [14.4 to 30.4] | 28 [20.2 to 37.9] | 26 [17.3 to 35.9] | 31 [19.9 to 43.4] | 36 [23.1 to 50.2] | 54 [46 to 61.4] | 49 [34.4 to 63.7]

3. Primary Outcome: The hSBA Geometric Mean Titers (GMTs) Against N.Meningitidis Serogroup B Strains
Description: The hSBA antibody titers in subjects, 24 to 36 months after completion of Bexsero® vaccination course according to different schedules in the parent study, are presented in terms of vaccine-group-specific GMTs, alongside with the corresponding antibody responses in age-matched vaccine-naïve subjects at baseline.
Time Frame: 24-36 months after booster dose in the parent study; baseline for vaccine-naïve subjects
Population: Analysis was done on FAS-persistence: All subjects in the Enrolled Set who provide an evaluable serum sample at Visit 1. The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | 2H3H511 | 3H5_11 | 68_11 | NAIVE 123 | 02_2_5 | NAIVE_4A | 02_6_10 | NAIVE_4B
Number analyzed (Participants) | 140 | 131 | 119 | 100 | 68 | 55 | 179 | 50
Titers
  H44/76: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 178 | 50
  H44/76 | 4.17 [3.4 to 5.13] | 4.48 [3.6 to 5.57] | 5.62 [4.48 to 7.04] | 2.79 [2.25 to 3.45] | 3.97 [2.99 to 5.28] | 2.33 [1.77 to 3.07] | 5.75 [4.78 to 6.91] | 1.93 [1.39 to 2.68]
  5/99: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  5/99 | 44 [32 to 60] | 52 [37 to 72] | 83 [58 to 117] | 1.15 [1.03 to 1.29] | 21 [14 to 33] | 1.2 [0.96 to 1.51] | 21 [16 to 28] | 1.38 [1.1 to 1.73]
  NZ98/254: number analyzed (Participants) | 140 | 131 | 119 | 100 | 67 | 55 | 179 | 50
  NZ98/254 | 3.48 [2.78 to 4.36] | 2.98 [2.35 to 3.78] | 4.86 [3.8 to 6.22] | 1.14 [1.06 to 1.22] | 2.81 [2.07 to 3.82] | 1.37 [1.17 to 1.61] | 4.57 [3.74 to 5.59] | 1.22 [1.06 to 1.41]
  M10713: number analyzed (Participants) | 127 | 111 | 109 | 93 | 65 | 53 | 173 | 49
  M10713 | 2.77 [2.06 to 3.71] | 3.03 [2.2 to 4.16] | 3.17 [2.3 to 4.38] | 3.3 [2.52 to 4.32] | 3.53 [2.38 to 5.25] | 4.26 [2.61 to 6.97] | 7.82 [6.04 to 10] | 6.95 [4.18 to 12]

4. Primary Outcome: The Geometric Mean Ratio (GMR) of hSBA GMTs Against N. Meningitidis Serogroup B, 24 to 36 Months Versus 1 Month After Completion of Bexsero® Vaccination Course According to Different Schedules in the Parent Study.
Description: The within-subjects GMR of GMTs at 24 to 36 months versus 1 month after completion of Bexsero® vaccination course according to different schedules vaccination in parent study are reported.
Time Frame: At Day 1 in this study over one month after the completion of the vaccination course in the parent study
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2H3H511 | 3H5_11 | 68_11 | 02_2_5 | 02_6_10
Number analyzed (Participants) | 137 | 130 | 118 | 68 | 176
Ratio
  H44/76: number analyzed (Participants) | 137 | 129 | 118 | 67 | 173
  H44/76 | 0.029 [0.023 to 0.036] | 0.022 [0.017 to 0.028] | 0.03 [0.023 to 0.038] | 0.028 [0.021 to 0.038] | 0.042 [0.035 to 0.052]
  5/99: number analyzed (Participants) | 136 | 130 | 118 | 66 | 176
  5/99 | 0.023 [0.017 to 0.03] | 0.031 [0.023 to 0.041] | 0.054 [0.04 to 0.073] | 0.045 [0.031 to 0.066] | 0.049 [0.038 to 0.063]
  NZ98/254: number analyzed (Participants) | 136 | 129 | 116 | 68 | 174
  NZ98/254 | 0.059 [0.047 to 0.074] | 0.038 [0.03 to 0.048] | 0.07 [0.055 to 0.09] | 0.061 [0.044 to 0.083] | 0.095 [0.077 to 0.12]
  M10713: number analyzed (Participants) | 105 | 84 | 78 | 61 | 160
  M10713 | 0.19 [0.13 to 0.28] | 0.16 [0.11 to 0.25] | 0.19 [0.12 to 0.29] | 0.17 [0.11 to 0.28] | 0.24 [0.17 to 0.32]

5. Primary Outcome: The Geometric Mean Ratio (GMR) of hSBA GMTs Against N. Meningitidis Serogroup B, 24 to 36 Months Versus Visit 1 in the Parent Study.
Description: The within-subjects GMR of GMTs at 24 to 36 months versus visit 1 in the vaccination course according to different schedules vaccination in the parent study are reported.
Time Frame: At Day 1 in this study over visit 1 in the vaccination course in the parent study
Population: Analysis was done on FAS-persistence: All subjects in the Enrolled Set who provide an evaluable serum sample at Visit 1.This outcome measure applies to only groups 02_2_5 & 02_6_10 as the GMRs were calculated at 24-36 months after completion of vaccination course in the parent study over subjects belonging to groups 02_2_5 & 02_6_10.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 02_2_5 | 02_6_10
Number analyzed (Participants) | 67 | 177
Ratio
  H44/76 | 1.88 [1.32 to 2.69] | 2.94 [2.33 to 3.71]
  5/99 | 20 [12 to 32] | 14 [10 to 20]
  NZ98/254 | 2.48 [1.76 to 3.49] | 3.06 [2.44 to 3.83]
  M10713: number analyzed (Participants) | 56 | 163
  M10713 | 0.89 [0.49 to 1.61] | 0.94 [0.64 to 1.37]

6. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥4 or ≥ 5 Against N.Meningitidis Serogroup B, After Receiving Bexsero® Booster Vaccination in This Study.
Description: The percentage of subjects with hSBA titers ≥ 4 against H44/76, 5/99 and NZ98/254 strains, and with hSBA titers ≥ 5 against M10713 strain, after receiving Bexsero® booster vaccination in this study (24 to 36 months after completion of vaccination course according to different schedules in parent study), alongside the corresponding response after the first dose of Bexsero® vaccine in age matched vaccine-naïve subjects.
Time Frame: At 24-36 months (Visit 1) and one month after booster vaccination (Day 31)
Population: Analysis was done on FAS - booster: All subjects in the Enrolled Set who receive a study vaccination and provide an evaluable serum sample at visit 2 (one month after the booster dose administration) and received all scheduled vaccinations in the parent study V72_28 (excluding naïve groups).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 96 | 87 | 76 | 32 | 91 | 96 | 55 | 50
Percentage of subjects
  H44/76 (pre-vacc.): number analyzed (Participants) | 92 | 87 | 75 | 31 | 91 | 96 | 55 | 50
  H44/76 (pre-vacc.) | 48 [37.3 to 58.5] | 51 [40.1 to 62.1] | 64 [52.1 to 74.8] | 39 [21.8 to 57.8] | 59 [48.5 to 69.5] | 39 [28.8 to 49] | 27 [16.1 to 41] | 20 [10 to 33.7]
  H44/76 (post-vacc.): number analyzed (Participants) | 96 | 87 | 75 | 32 | 91 | 96 | 55 | 50
  H44/76 (post-vacc.) | 99 [94.3 to 99.97] | 100 [95.8 to 100] | 100 [95.2 to 100] | 97 [83.8 to 99.92] | 99 [94 to 99.97] | 95 [88.3 to 98.3] | 91 [80 to 97] | 80 [66.3 to 90]
  5/99 (pre-vacc.): number analyzed (Participants) | 92 | 87 | 76 | 31 | 91 | 96 | 55 | 50
  5/99 (pre-vacc.) | 84 [74.5 to 90.6] | 91 [82.7 to 95.9] | 95 [87.1 to 98.5] | 74 [55.4 to 88.1] | 86 [76.8 to 92.2] | 3 [0.6 to 8.9] | 4 [0.44 to 12.5] | 8 [2.2 to 19.2]
  5/99 (post-vacc.) | 99 [94.3 to 99.97] | 99 [93.8 to 99.97] | 97 [90.8 to 99.68] | 100 [89.1 to 100] | 100 [96 to 100] | 88 [79.2 to 93.4] | 93 [82.4 to 98] | 80 [66.3 to 90]
  NZ98/254 (pre-vacc.): number analyzed (Participants) | 92 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/254 (pre-vacc.) | 45 [34.2 to 55.3] | 42 [31.3 to 53] | 52 [40.2 to 63.7] | 25 [11.5 to 43.4] | 47 [36.7 to 58] | 2 [0.25 to 7.3] | 7 [2.1 to 17.9] | 6 [1.3 to 16.5]
  NZ98/254 (post-vacc.): number analyzed (Participants) | 96 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/254 (post-vacc.) | 99 [94.3 to 99.97] | 100 [95.8 to 100] | 100 [95.2 to 100] | 100 [89.1 to 100] | 100 [96 to 100] | 78 [68.5 to 85.9] | 85 [72.9 to 93.4] | 70 [55.4 to 82.1]
  M10713 (pre-vacc.): number analyzed (Participants) | 78 | 68 | 65 | 29 | 87 | 84 | 49 | 46
  M10713 (pre-vacc.) | 36 [25.3 to 47.6] | 35 [24.1 to 47.8] | 45 [32.3 to 57.5] | 21 [8 to 39.7] | 63 [52.2 to 73.3] | 39 [28.8 to 50.5] | 41 [27 to 55.8] | 59 [43.2 to 73]
  M10713 (post-vacc.): number analyzed (Participants) | 88 | 79 | 67 | 30 | 89 | 88 | 51 | 47
  M10713 (post-vacc.) | 70 [59.8 to 79.7] | 81 [70.6 to 89] | 97 [89.6 to 99.64] | 97 [77.9 to 99.2] | 96 [88.9 to 98.8] | 47 [35.9 to 57.5] | 59 [44.2 to 72.4] | 60 [44.3 to 73.6]

7. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥ 8 Against N.Meningitidis serogroupB, After Receiving Bexsero® Booster Vaccination in This Study.
Description: The percentage of subjects with hSBA titers ≥ 8, after receiving Bexsero® booster vaccination in this study (24 to 36 months after completion of vaccination course according to different schedules in parent study) alongside the corresponding response after the first dose of Bexsero® vaccine in age matched vaccine-naïve subjects.
Time Frame: At 24-36 months (Visit 1) and one month after booster vaccination (Day 31)
Population: Analysis was done on FAS-booster:All subjects in the Enrolled Set who receive a study vaccination & provide an evaluable serum sample at visit 2(1 month post booster dose) & received all scheduled vaccinations in V72_28 (excluding naïve groups).The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 96 | 87 | 76 | 32 | 91 | 96 | 55 | 50
Percentage of subjects
  H44/76 (pre-vacc.): number analyzed (Participants) | 92 | 86 | 75 | 31 | 91 | 96 | 55 | 50
  H44/76 (pre-vacc.) | 26 [17.5 to 36.3] | 31 [21.8 to 42.3] | 33 [22.9 to 45.2] | 19 [7.5 to 37.5] | 30 [20.5 to 40.2] | 18 [10.7 to 26.8] | 16 [7.8 to 28.8] | 10 [3.3 to 21.8]
  H44/76 (post-vacc.): number analyzed (Participants) | 96 | 86 | 75 | 32 | 91 | 96 | 55 | 50
  H44/76 (post-vacc.) | 97 [91.1 to 99.4] | 98 [91.9 to 99.72] | 99 [92.8 to 99.97] | 97 [83.8 to 99.92] | 97 [90.7 to 99.3] | 68 [57.4 to 76.9] | 71 [57.1 to 82.4] | 60 [45.2 to 73.6]
  5/99 (pre-vacc.): number analyzed (Participants) | 92 | 87 | 76 | 31 | 91 | 96 | 55 | 50
  5/99 (pre-vacc.) | 79 [69.6 to 87.1] | 85 [75.8 to 91.8] | 91 [81.9 to 96.2] | 71 [52 to 85.8] | 68 [57.5 to 77.5] | 2 [0.25 to 7.3] | 4 [0.44 to 12.5] | 6 [1.3 to 16.5]
  5/99 (post-vacc.) | 99 [94.3 to 99.97] | 99 [93.8 to 99.97] | 97 [90.8 to 99.68] | 100 [89.1 to 100] | 100 [96 to 100] | 77 [67.4 to 85] | 78 [65 to 88.2] | 60 [45.2 to 73.6]
  NZ98/254 (pre-vacc.): number analyzed (Participants) | 92 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/254 (pre-vacc.) | 22 [13.8 to 31.6] | 19 [11 to 28.4] | 28 [18.2 to 39.6] | 13 [3.5 to 29] | 26 [17.7 to 36.7] | 0 [0 to 3.8] | 2 [0.05 to 9.9] | 0 [0 to 7.1]
  NZ98/54 (post-vacc.): number analyzed (Participants) | 96 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/54 (post-vacc.) | 97 [91.1 to 99.4] | 98 [91.9 to 99.72] | 100 [95.2 to 100] | 97 [83.8 to 99.92] | 97 [90.7 to 99.3] | 34 [25 to 44.8] | 54 [39.6 to 67.4] | 40 [26.4 to 54.8]
  M10713 (pre-vacc.): number analyzed (Participants) | 78 | 68 | 65 | 29 | 87 | 84 | 49 | 46
  M10713 (pre-vacc.) | 28 [18.6 to 39.5] | 22 [12.9 to 33.8] | 34 [22.6 to 46.6] | 17 [5.8 to 35.8] | 55 [44.1 to 65.9] | 27 [18.2 to 38.2] | 39 [25.2 to 53.8] | 52 [36.9 to 67.1]
  M10713 (post-vacc.): number analyzed (Participants) | 88 | 79 | 67 | 30 | 89 | 88 | 51 | 47
  M10713 (post-vacc.) | 64 [52.7 to 73.6] | 71 [59.6 to 80.6] | 94 [85.4 to 98.3] | 90 [73.5 to 97.9] | 92 [84.5 to 96.8] | 34 [24.3 to 45] | 51 [36.6 to 65.2] | 57 [42.2 to 71.7]

8. Secondary Outcome: Percentage of Subjects With Four-fold Rise in hSBA Titers, After Receiving Bexsero® Vaccination in This Study.
Description: The percentage of subjects with a four-fold rise in hSBA titers 1 month after receiving Bexsero® booster vaccination in this study to pre vaccination at visit 1 (24 to 36 months after completion of vaccination course according to different schedules in parent study) alongside the corresponding response after the first dose of Bexsero® vaccine in age matched vaccine-naïve subjects.
Time Frame: One month after booster vaccination (day 31)/24-36 months (Visit 1)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 92 | 87 | 76 | 32 | 91 | 96 | 55 | 50
Percentage of subjects
  H44/76 (Day 31/PRE): number analyzed (Participants) | 92 | 86 | 75 | 31 | 91 | 96 | 55 | 50
  H44/76 (Day 31/PRE) | 95 [87.8 to 98.2] | 95 [88.5 to 98.7] | 97 [90.7 to 99.68] | 94 [78.6 to 99.2] | 97 [90.7 to 99.3] | 43 [32.7 to 53.2] | 53 [38.8 to 66.3] | 46 [31.8 to 60.7]
  5/99 (Day 31/PRE): number analyzed (Participants) | 92 | 87 | 76 | 31 | 91 | 96 | 55 | 50
  5/99 (Day 31/PRE) | 98 [92.4 to 99.74] | 98 [91.9 to 99.72] | 95 [87.1 to 98.5] | 100 [88.8 to 100] | 98 [92.3 to 99.73] | 77 [67.4 to 85] | 76 [63 to 86.8] | 60 [45.2 to 73.6]
  NZ98/254 (Day 31/PRE): number analyzed (Participants) | 92 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/254 (Day 31/PRE) | 92 [84.9 to 96.9] | 95 [88.5 to 98.7] | 93 [85.1 to 97.8] | 94 [79.2 to 99.2] | 86 [76.8 to 92.2] | 34 [25 to 44.8] | 54 [39.6 to 67.4] | 40 [26.4 to 54.8]
  M10713 (Day 31/PRE): number analyzed (Participants) | 78 | 68 | 65 | 29 | 87 | 84 | 49 | 46
  M10713 (Day 31/PRE) | 41 [30 to 52.7] | 50 [37.6 to 62.4] | 68 [54.9 to 78.8] | 72 [52.8 to 87.3] | 53 [41.9 to 63.7] | 11 [5 to 19.4] | 20 [10.2 to 34.3] | 13 [4.9 to 26.3]

9. Secondary Outcome: Percentage of Subjects With Four-fold Rise in hSBA Titers, One Month After Receiving Bexsero® Vaccination in This Study
Description: The percentage of subjects with a four-fold rise in hSBA titers one month after receiving Bexsero® booster vaccination (visit 2) in this study to post primary visit in the parent study V72_28(1 month after last vaccination in the parent study) alongside the corresponding response after the first dose of Bexsero® vaccine in age matched vaccine-naïve subjects.
Time Frame: From post primary visit in the parent study to visit 2 in this extension study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V
Number analyzed (Participants) | 94 | 86 | 76 | 32 | 89
Percentage of subjects
  H44/76: number analyzed (Participants) | 94 | 84 | 75 | 32 | 88
  H44/76 | 5 [1.7 to 12.0] | 5 [1.3 to 11.7] | 13 [6.6 to 23.2] | 22 [9.3 to 40.0] | 17 [9.9 to 26.6]
  5/99: number analyzed (Participants) | 93 | 86 | 76 | 32 | 89
  5/99 | 19 [11.9 to 28.9] | 27 [17.8 to 37.4] | 37 [26.1 to 48.7] | 66 [46.8 to 81.4] | 72 [61.4 to 80.9]
  NZ98/254: number analyzed (Participants) | 93 | 84 | 73 | 32 | 88
  NZ98/254 | 25 [16.4 to 34.8] | 15 [8.5 to 25.0] | 27 [17.6 to 39.1] | 13 [3.5 to 29.0] | 18 [10.8 to 27.8]
  M10713: number analyzed (Participants) | 74 | 57 | 50 | 29 | 81
  M10713 | 15 [7.7 to 25.0] | 21 [11.4 to 33.9] | 24 [13.1 to 38.2] | 21 [8.0 to 39.7] | 11 [5.2 to 20.0]

10. Secondary Outcome: Percentage of Subjects With Four-fold Rise in hSBA Titers, One Month After Receiving Bexsero® Vaccination in This Study.
Description: The percentage of subjects with a four-fold rise in hSBA titers one month after receiving Bexsero® booster vaccination in this study to pre primary visit in parent study V72_28 (Visit 1). This outcome measure was analysed only for subjects belonging to groups 02_2_5_V and 02_6_10_V
Time Frame: From pre primary visit in the parent study (Visit 1) to visit 2 in this extension study
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 02_2_5_V | 02_6_10_V
Number analyzed (Participants) | 32 | 91
Percentage of subjects
  H44/76 | 97 [83.8 to 99.92] | 96 [89.1 to 98.8]
  5/99: number analyzed (Participants) | 32 | 90
  5/99 | 100 [89.1 to 100.0] | 100 [96.0 to 100.0]
  NZ98/254: number analyzed (Participants) | 31 | 90
  NZ98/254 | 94 [78.6 to 99.2] | 97 [90.6 to 99.3]
  M10713: number analyzed (Participants) | 27 | 82
  M10713 | 67 [46.0 to 83.5] | 55 [43.5 to 65.9]

11. Secondary Outcome: The GMTs Against N.Meningitidis Serogroup B, One Month After Receiving Bexsero® Booster Vaccination in the Present Study.
Description: The hSBA antibody titers in subjects after receiving Bexsero® booster vaccination in this study (24 to 36 months after completion of vaccination course according to different schedules in parent study) alongside the corresponding response after the 1st dose of Bexsero® vaccine in age matched vaccine-naïve subjects in terms of GMTs.
Time Frame: At Visit 1 and one month post booster vaccination (Day 31)
Population: Analysis was done on FAS-Booster:All subjects in the Enrolled Set who receive a study vaccination & provide an evaluable serum sample at visit 2(1 month post booster dose) & received all scheduled vaccinations in V72_28(excluding naïve groups).The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 96 | 87 | 76 | 32 | 91 | 96 | 55 | 50
Titers | 3.91 [3.01 to 5.08] | 4.84 [3.66 to 6.41] | 6.21 [4.65 to 8.31] | 3.14 [2.08 to 4.75] | 6.15 [4.77 to 7.93] | 2.82 [2.26 to 3.5] | 2.33 [1.77 to 3.07] | 1.93 [1.39 to 2.68]

12. Secondary Outcome: The Geometric Mean Ratio (GMR) of hSBA Titers, One Month After Receiving Bexsero® Booster Vaccination in the Present Study.
Description: The within-subjects GMR of hSBA antibody titers (one month post booster vaccination versus pre vaccination) after Bexsero® booster vaccination in this study (24 to 36 months after completion of vaccination course according to different schedules in parent study) alongside the within-subject GMR for the 1st dose of rMenB+OMV NZ vaccination of age matched naïve subjects.
Time Frame: At Day 31 versus Day 1
Population: Analysis was done on FAS-Booster:All subjects in the Enrolled Set who receive a study vaccination & provide an evaluable serum sample at visit 2 (1 month post booster dose) & received all scheduled vaccinations in V72_28 (excluding naïve groups). The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 92 | 87 | 76 | 32 | 91 | 96 | 55 | 50
Ratio
  H44/76 (Day 31/PRE): number analyzed (Participants) | 92 | 86 | 75 | 31 | 91 | 96 | 55 | 50
  H44/76 (Day 31/PRE) | 41 [30 to 55] | 43 [31 to 59] | 46 [33 to 65] | 50 [31 to 80] | 42 [31 to 56] | 4.81 [3.81 to 6.07] | 7.08 [5.07 to 9.88] | 6.87 [4.62 to 10]
  5/99 (Day 31/PRE): number analyzed (Participants) | 92 | 87 | 76 | 31 | 91 | 96 | 55 | 50
  5/99 (Day 31/PRE) | 75 [54 to 104] | 67 [47 to 96] | 41 [29 to 60] | 160 [95 to 270] | 135 [98 to 186] | 34 [24 to 46] | 22 [15 to 34] | 14 [9.11 to 23]
  NZ98/254 (Day 31/PRE): number analyzed (Participants) | 92 | 86 | 75 | 32 | 91 | 96 | 54 | 50
  NZ98/254 (Day 31/PRE) | 28 [20 to 38] | 29 [21 to 41] | 27 [19 to 39] | 24 [15 to 40] | 18 [13 to 25] | 6.07 [4.97 to 7.41] | 9.58 [6.8 to 13] | 7.01 [4.54 to 11]
  M10713 (Day 31/PRE): number analyzed (Participants) | 78 | 68 | 65 | 29 | 87 | 84 | 49 | 46
  M10713 (Day 31/PRE) | 4.07 [2.8 to 5.91] | 5.65 [3.77 to 8.47] | 11 [7.15 to 16] | 13 [7.29 to 23] | 6.85 [4.86 to 9.66] | 1.38 [1.01 to 1.88] | 2.06 [1.36 to 3.12] | 1.55 [1.1 to 2.18]

13. Secondary Outcome: The Geometric Mean Ratio (GMR) of hSBA Titers, One Month After Receiving Bexsero® Booster Vaccination in the Present Study.
Description: The within-subjects GMR of hSBA antibody titers (one month post booster vaccination in this study versus 1 month post last vaccination visit (post-primary vaccination visit) in parent study V72_28.
Time Frame: Visit 2 (day 31 in extension study) versus post primary vaccination visit in parent study
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- 2H3H511_V: In the parent study V72_28 (NCT01894919), subjects received three primary doses and one booster dose of Bexsero® vaccine at 2.5, 3.5 and 5 months and at 11 months of age, respectively. The subjects in this group received a 5th dose of Bexsero® vaccine in the present study.
- 3H5_11_V: In the parent study V72_28 (NCT01894919), subjects received two primary doses and one booster dose of Bexsero® vaccine at 3.5 and 5 months and at 11 months of age, respectively. These subjects received a 4th dose of Bexsero® vaccine in the present study.
- 68_11_V: In the parent study V72_28 (NCT01894919), subjects received two primary doses and one booster dose of Bexsero® vaccine at 6 and 8 months and at 11 months of age, respectively. These subjects received a 4th dose of Bexsero® vaccine in the present study.
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V
Number analyzed (Participants) | 94 | 86 | 76
Ratio
  H44/76: number analyzed (Participants) | 94 | 84 | 75
  H44/76 | 1.06 [0.82 to 1.38] | 0.90 [0.68 to 1.20] | 1.37 [1.02 to 1.84]
  5/99: number analyzed (Participants) | 93 | 86 | 76
  5/99 | 1.60 [1.20 to 2.13] | 2.07 [1.52 to 2.82] | 2.33 [1.69 to 3.20]
  NZ98/254: number analyzed (Participants) | 93 | 84 | 73
  NZ98/254 | 1.66 [1.25 to 2.20] | 1.10 [0.81 to 1.49] | 1.75 [1.28 to 2.41]
  M10713: number analyzed (Participants) | 74 | 57 | 50
  M10713 | 1.01 [0.65 to 1.58] | 1.37 [0.82 to 2.29] | 2.35 [1.37 to 4.02]

14. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥ 4 or ≥ 5, After Receiving Two Catch up Doses of Bexsero® Vaccination
Description: The percentage of vaccine-naïve subjects with hSBA titers ≥ 4 against H44/76, 5/99 and NZ98/254 strains, and ≥ 5 against M10713 strain, one month after receiving two catch up doses of Bexsero® booster vaccination in this study.
Time Frame: At Baseline and One month post second vaccination (Day 61)
Population: Analysis was done on FAS-catch-up population: All subjects in the Enrolled Set who receive at least one study vaccination and provide evaluable serum samples whose assay results are available on at least one post-baseline visit (visit 1 or visit 2).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 98 | 54 | 49
Percentage of subjects
  H44/76 (baseline) | 38 [28.2 to 48.1] | 26 [15 to 39.7] | 20 [10.2 to 34.3]
  H44/76 (Day 61) | 100 [96.3 to 100] | 98 [90.1 to 99.95] | 100 [92.7 to 100]
  5/99 (baseline) | 3 [0.6 to 8.7] | 4 [0.45 to 12.7] | 6 [1.3 to 16.9]
  5/99 (Day 61) | 100 [96.3 to 100] | 100 [93.4 to 100] | 100 [92.7 to 100]
  NZ98/254 (baseline): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (baseline) | 2 [0.25 to 7.2] | 7 [2.1 to 17.9] | 6 [1.3 to 17.2]
  NZ98/254 (Day 61): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (Day 61) | 100 [96.3 to 100] | 100 [93.4 to 100] | 100 [92.6 to 100]
  M10713 (baseline): number analyzed (Participants) | 87 | 50 | 49
  M10713 (baseline) | 34 [24.6 to 45.4] | 40 [26.4 to 54.8] | 55 [40.2 to 69.3]
  M10713 (Day 61): number analyzed (Participants) | 91 | 52 | 49
  M10713 (Day 61) | 75 [64.5 to 83.3] | 69 [54.9 to 81.3] | 76 [61.1 to 86.7]

15. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥ 8 , After Receiving Two Catch up Doses of Bexsero® Vaccination.
Description: The percentage of vaccine-naïve subjects with hSBA titers ≥8, one month after receiving two catch up doses of Bexsero® booster vaccination in this study are reported.
Time Frame: At Baseline and One month post second vaccination (Day 61)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 98 | 54 | 49
Percentage of subjects
  H44/76 (baseline) | 17 [10.4 to 26.3] | 15 [6.6 to 27.1] | 10 [3.4 to 22.2]
  H44/76 (Day 61) | 99 [94.4 to 99.97] | 96 [87.3 to 99.55] | 98 [89.1 to 99.95]
  5/99 (baseline) | 2 [0.25 to 7.2] | 4 [0.45 to 12.7] | 4 [0.5 to 14]
  5/99 (Day 61) | 100 [96.3 to 100] | 100 [93.4 to 100] | 98 [89.1 to 99.95]
  NZ98/254 (baseline): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (baseline) | 0 [0 to 3.7] | 2 [0.05 to 9.9] | 0 [0 to 7.4]
  NZ98/254 (Day 61): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (Day 61) | 96 [89.9 to 98.9] | 93 [82.1 to 97.9] | 94 [82.8 to 98.7]
  M10713 (baseline): number analyzed (Participants) | 87 | 50 | 49
  M10713 (baseline) | 25 [16.6 to 35.7] | 38 [24.7 to 52.8] | 49 [34.4 to 63.7]
  M10713 (Day 61): number analyzed (Participants) | 91 | 52 | 49
  M10713 (Day 61) | 65 [54.1 to 74.6] | 63 [49 to 76.4] | 69 [54.6 to 81.7]

16. Secondary Outcome: Percentage of Subjects With Four-fold Rise in hSBA Titers, After Receiving Two Catch up Doses of Bexsero® Vaccination.
Description: The percentage of vaccine-naïve subjects with a four-fold rise in hSBA titers from baseline, one month after receiving two catch up doses of Bexsero® booster vaccination in comparison to prevaccination in this study are reported.
Time Frame: One month post second vaccination (Day 61)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 98 | 54 | 49
Percentage of subjects
  H44/76 | 94 [87.1 to 97.7] | 89 [77.4 to 95.8] | 94 [83.1 to 98.7]
  5/99 | 100 [96.3 to 100] | 100 [93.4 to 100] | 98 [89.1 to 99.95]
  NZ98/254: number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 | 94 [87.1 to 97.7] | 91 [79.7 to 96.9] | 94 [82.8 to 98.7]
  M10713: number analyzed (Participants) | 87 | 50 | 49
  M10713 | 37 [26.7 to 47.8] | 28 [16.2 to 42.5] | 22 [11.8 to 36.6]

17. Secondary Outcome: The GMTs in Subjects Who Received Two Catch up Doses of Bexsero® Vaccination.
Description: The hSBA antibody titers in vaccine-naïve subjects , after receiving two catch up doses of Bexsero® vaccination in this study, are reported in terms of GMTs.
Time Frame: At Baseline and One month post second vaccination (Day 61)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 98 | 54 | 49
Titers
  H44/76 (baseline) | 2.3 [1.75 to 3.01] | 2.15 [1.55 to 3] | 1.56 [1.11 to 2.2]
  H44/76 (Day 61) | 107 [84 to 135] | 74 [56 to 99] | 63 [47 to 85]
  5/99 (baseline) | 1.13 [0.94 to 1.36] | 1.13 [0.9 to 1.41] | 1.31 [1.04 to 1.65]
  5/99 (Day 61) | 631 [503 to 792] | 421 [319 to 555] | 317 [238 to 423]
  NZ98/254 (baseline): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (baseline) | 1.11 [0.98 to 1.26] | 1.34 [1.15 to 1.56] | 1.2 [1.02 to 1.4]
  NZ98/254 (Day 61): number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 (Day 61) | 34 [27 to 42] | 37 [28 to 49] | 34 [26 to 46]
  M10713 (baseline): number analyzed (Participants) | 87 | 50 | 49
  M10713 (baseline) | 2.9 [1.94 to 4.34] | 4.12 [2.54 to 6.69] | 6.4 [3.91 to 10]
  M10713 (Day 61): number analyzed (Participants) | 91 | 52 | 49
  M10713 (Day 61) | 12 [7.57 to 18] | 11 [6.87 to 19] | 14 [8.34 to 24]

18. Secondary Outcome: The GMRs of hSBA Titers After Two Catch up Doses of Bexsero® Vaccination Versus hSBA Titers at Baseline.
Description: The within-subject GMRs of hSBA titers at one month after receiving the second catch up dose to hSBA titers at baseline, for naïve subjects who received two catch up doses of Bexsero® vaccination in this study are reported.
Time Frame: At one month after receiving second vaccination (Day 61) versus baseline (Day 1)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 98 | 54 | 49
Ratio
  H44/76 | 46 [34 to 63] | 34 [24 to 50] | 41 [27 to 60]
  5/99 | 558 [423 to 737] | 373 [266 to 524] | 242 [171 to 344]
  NZ98/254: number analyzed (Participants) | 98 | 54 | 48
  NZ98/254 | 30 [24 to 39] | 27 [20 to 37] | 29 [21 to 39]
  M10713: number analyzed (Participants) | 87 | 50 | 49
  M10713 | 3.86 [2.62 to 5.69] | 2.93 [1.84 to 4.67] | 2.2 [1.37 to 3.53]

19. Secondary Outcome: Number of Subjects (35 Months to 7 Years of Age) Reporting Solicited Local and Systemic Adverse Events After Receiving Bexsero® Booster Vaccine.
Description: The number of subjects (35 months to 7 years of age) with solicited local and systemic adverse events after receiving Bexsero® booster vaccine in the present study.
Time Frame: From day 1 (6 hr) through day 7 after vaccination
Population: Analysis was done on solicited safety set: All subjects in the Exposed Set with solicited adverse event data
Measure: Number; unit: Subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V
Number analyzed (Participants) | 97 | 89 | 80 | 32
Subjects
  Any local AEs | 87 | 81 | 73 | 31
  Erythema | 60 | 63 | 42 | 22
  Induration | 48 | 48 | 33 | 15
  Swelling | 49 | 50 | 37 | 20
  Tenderness | 84 | 80 | 71 | 31
  Any systemic AEs | 66 | 63 | 54 | 18
  Change in eating habits | 31 | 32 | 30 | 5
  Diarrhea | 4 | 8 | 5 | 0
  Irritability | 54 | 52 | 46 | 9
  Persistent Crying | 31 | 24 | 25 | 4
  Rash | 13 | 1 | 3 | 5
  Sleepiness | 28 | 23 | 26 | 5
  Vomiting | 5 | 5 | 2 | 1
  Fever (>38.0° C) | 17 | 18 | 11 | 2
  Medically-Attended Fever | 1 | 0 | 2 | 0
  Prevention of Pain and/or Fever | 23 | 14 | 15 | 1
  Treatment of Pain and/or Fever | 38 | 39 | 41 | 13

20. Secondary Outcome: Number of Newly Recruited Subjects (Aged 35 Months to 7 Years) Reporting Solicited Local and Systemic Adverse Events After Receiving Catch-up Doses of Bexsero® Vaccine.
Description: The number of newly recruited subjects (aged 35 months to 7 years) reporting solicited local and systemic adverse events after receiving two catch-up doses of Bexsero® vaccine in the present study.
Time Frame: From day 1 (6 hr) through day 7 after vaccination
Population: Analysis was done on solicited safety set: All subjects in the Exposed Set with solicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | NAIVE 123 | NAIVE_4A
Number analyzed (Participants) | 100 | 55
Subjects
  Any local AEs (1st vacc.) | 88 | 55
  Erythema (1st vacc.) | 54 | 28
  Induration (1st vacc.) | 38 | 17
  Swelling (1st vacc.) | 40 | 24
  Tenderness (1st vacc.) | 87 | 55
  Any systemic AEs (1st vacc.) | 64 | 24
  Change in Eating Habits (1st vacc.) | 31 | 5
  Diarrhea (1st vacc.) | 4 | 3
  Irritability (1st vacc.) | 40 | 16
  Persistent Crying (1st vacc.) | 15 | 4
  Rash (1st vacc.) | 5 | 3
  Sleepiness (1st vacc.) | 18 | 9
  Vomiting (1st vacc.) | 7 | 2
  Fever (>38.0° C) (1st vacc.) | 15 | 2
  Medically-Attended Fever (1st vacc.) | 1 | 0
  Prevention of Pain/Fever (1st vacc.) | 18 | 3
  Treatment of Pain/Fever (1st vacc.): number analyzed (Participants) | 99 | 55
  Treatment of Pain/Fever (1st vacc.) | 41 | 22
  Any local AEs (2nd vacc.): number analyzed (Participants) | 99 | 55
  Any local AEs (2nd vacc.) | 79 | 51
  Erythema (2nd vacc.): number analyzed (Participants) | 99 | 55
  Erythema (2nd vacc.) | 44 | 32
  Induration (2nd vacc.): number analyzed (Participants) | 99 | 55
  Induration (2nd vacc.) | 29 | 22
  Swelling (2nd vacc.): number analyzed (Participants) | 99 | 55
  Swelling (2nd vacc.) | 32 | 25
  Tenderness (2nd vacc.): number analyzed (Participants) | 99 | 55
  Tenderness (2nd vacc.) | 77 | 51
  Any systemic AEs (2nd vacc.): number analyzed (Participants) | 99 | 55
  Any systemic AEs (2nd vacc.) | 46 | 18
  Change in Eating Habits (2nd vacc.): number analyzed (Participants) | 99 | 55
  Change in Eating Habits (2nd vacc.) | 15 | 9
  Diarrhea (2nd vacc.): number analyzed (Participants) | 99 | 55
  Diarrhea (2nd vacc.) | 2 | 3
  Irritability (2nd vacc.): number analyzed (Participants) | 99 | 55
  Irritability (2nd vacc.) | 25 | 11
  Persistent Crying (2nd vacc.): number analyzed (Participants) | 99 | 55
  Persistent Crying (2nd vacc.) | 13 | 6
  Rash (2nd vacc.): number analyzed (Participants) | 99 | 55
  Rash (2nd vacc.) | 2 | 1
  Sleepiness (2nd vacc.): number analyzed (Participants) | 99 | 55
  Sleepiness (2nd vacc.) | 12 | 5
  Vomiting (2nd vacc.): number analyzed (Participants) | 99 | 55
  Vomiting (2nd vacc.) | 4 | 2
  Fever (>38.0° C) (2nd vacc.): number analyzed (Participants) | 99 | 55
  Fever (>38.0° C) (2nd vacc.) | 12 | 3
  Medically-Attended Fever (2nd vacc.): number analyzed (Participants) | 99 | 55
  Medically-Attended Fever (2nd vacc.) | 0 | 1
  Prevention of Pain/Fever (2nd vacc.): number analyzed (Participants) | 99 | 55
  Prevention of Pain/Fever (2nd vacc.) | 21 | 4
  Treatment of Pain/Fever (2nd vacc.): number analyzed (Participants) | 99 | 55
  Treatment of Pain/Fever (2nd vacc.) | 30 | 13

21. Secondary Outcome: Number of Subjects (8 to 12 Years of Age) Reporting Solicited Local and Systemic Adverse Events After Receiving Bexsero® Booster Vaccine.
Description: Number of subjects (8 to 12 years of age) reporting solicited local and systemic adverse events after receiving Bexsero® booster vaccine.
Time Frame: From day 1 (6 hr) through day 7 after vaccination
Population: Analysis was done on solicited safety set: All subjects in the Exposed Set with solicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | 02_6_10_V
Number analyzed (Participants) | 91
Subjects
  Any local AEs | 85
  Erythema | 57
  Induration | 44
  Swelling | 52
  Pain: number analyzed (Participants) | 90
  Pain | 84
  Any systemic AEs | 57
  Arthralgia: number analyzed (Participants) | 90
  Arthralgia | 18
  Chills: number analyzed (Participants) | 90
  Chills | 23
  Headache: number analyzed (Participants) | 90
  Headache | 27
  Malaise: number analyzed (Participants) | 90
  Malaise | 35
  Myalgia: number analyzed (Participants) | 90
  Myalgia | 24
  Nausea: number analyzed (Participants) | 90
  Nausea | 12
  Rash: number analyzed (Participants) | 90
  Rash | 10
  Fever (>38.0° C) | 10
  Medically-Attended Fever | 0
  Prevention of Pain and/or Fever: number analyzed (Participants) | 90
  Prevention of Pain and/or Fever | 12
  Treatment of Pain and/or Fever | 47

22. Secondary Outcome: Number of Newly Recruited naïve Subjects (Aged 8 to 12 Years of Age) Solicited Local and Systemic Adverse Events After Receiving Bexsero® Vaccine.
Description: The number newly recruited naïve subjects (aged 8 to12 years of age) reporting solicited local and systemic adverse events after receiving two catch-up doses of Bexsero® vaccine in the present study.
Time Frame: From day 1(6 hr) through day 7 after vaccination
Population: Analysis was done on solicited safety set: All subjects in the Exposed Set with solicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | NAIVE_4B
Number analyzed (Participants) | 50
Subjects
  Any local AEs (1st vacc.) | 49
  Erythema (1st vacc.) | 31
  Induration (1st vacc.) | 19
  Swelling (1st vacc.) | 29
  Pain (1st vacc.): number analyzed (Participants) | 49
  Pain (1st vacc.) | 47
  Any systemic AEs (1st vacc.) | 24
  Arthralgia (1st vacc.): number analyzed (Participants) | 49
  Arthralgia (1st vacc.) | 6
  Chills (1st vacc.): number analyzed (Participants) | 49
  Chills (1st vacc.) | 4
  Headache (1st vacc.): number analyzed (Participants) | 49
  Headache (1st vacc.) | 15
  Malaise (1st vacc.): number analyzed (Participants) | 49
  Malaise (1st vacc.) | 7
  Myalgia (1st vacc.): number analyzed (Participants) | 49
  Myalgia (1st vacc.) | 12
  Nausea (1st vacc.): number analyzed (Participants) | 49
  Nausea (1st vacc.) | 5
  Rash (1st vacc.) | 1
  Fever (>38.0° C) (1st vacc.) | 3
  Medically-Attended Fever (1st vacc.) | 0
  Prevention of Pain and/or Fever (1st vacc.) | 2
  Treatment of Pain and/or Fever (1st vacc.) | 21
  Any local AEs (2nd vacc.) | 43
  Erythema (2nd vacc.) | 21
  Induration (2nd vacc.) | 17
  Swelling (2nd vacc.) | 21
  Pain (2nd vacc.) | 41
  Any systemic AEs (2nd vacc.) | 25
  Arthralgia (2nd vacc.) | 3
  Chills (2nd vacc.) | 5
  Headache (2nd vacc.) | 10
  Malaise (2nd vacc.) | 13
  Myalgia (2nd vacc.) | 8
  Nausea (2nd vacc.) | 4
  Rash (2nd vacc.) | 3
  Fever (>38.0° C) (2nd vacc.) | 1
  Medically-Attended Fever (2nd vacc.) | 0
  Prevention of Pain and/or Fever (2nd vacc.) | 3
  Treatment of Pain and/or Fever (2nd vacc.) | 12

23. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving Bexsero® Vaccination.
Description: The number of subjects reporting unsolicited adverse events after receiving Bexsero® booster vaccination (24 to 36 months after completion of vaccination course according to different schedules in parent study) or two cach up schedule of Bexsero® vaccine is reported.
Time Frame: From day 1 through day 7 after any vaccination
Population: Analysis was done on unsolicited safety set: All subjects in the Exposed Set with unsolicited adverse event data.
Measure: Number; unit: Subjects
Groups:
- 3H5_11_V: In the parent study V72_28 (NCT01339923), subjects received three primary doses and one booster dose of Bexsero® vaccine at 2.5, 3.5 and 5 months and at 11 months of age, respectively. The subjects in this group received a 5th dose of Bexsero® vaccine in the present study.
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 96 | 89 | 78 | 32 | 91 | 100 | 55 | 50
Subjects
  Any AEs | 26 | 19 | 26 | 9 | 14 | 43 | 25 | 12
  Possibly or Probably Related AEs | 9 | 7 | 10 | 6 | 11 | 12 | 10 | 6
  AEs leading to Premature Withdrawal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

24. Secondary Outcome: Number of Subjects Reporting Unsolicited Serious Adverse Events (SAEs), Medically Attended AEs and AEs Leading to Withdrawal for Entire Study Period.
Description: The number of subjects reporting unsolicited SAEs, medically attended AEs and AEs leading to withdrawal after receiving Bexsero® booster vaccination (24 to 36 months after completion of vaccination course according to different schedules in the parent study) or two catch-up schedule of Bexsero® vaccine is reported.
Time Frame: Throughout the entire study period (up to 2 months)
Population: Analysis was done on unsolicited safety set: All subjects in the Exposed Set with unsolicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
Number analyzed (Participants) | 96 | 89 | 78 | 32 | 91 | 100 | 55 | 50
Subjects
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Possibly or probably related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs were collected from Day 1 (30 minutes) throughout Day 7; SAEs were collected throughout the entire study period (up to 2 months)
Description: Subjects in the 2H3H511_NV Group, 3H5_11_NV Group, 68_11_NV Group, 02_2_5_NV Group and 02_6_10_NV Group were only evaluated for antibody persistence and hence not included in the safety analysis.
Groups:
- 02_2_5_V; 02_6_10_V: In the parent study V72_28 (NCT01894919), these subjects received two catch-up doses of Bexsero® vaccine, two months apart. These subjects received a 3rd dose of Bexsero® vaccine in the present study.
Arm/Group | 2H3H511_V | 3H5_11_V | 68_11_V | 02_2_5_V | 02_6_10_V | NAIVE 123 | NAIVE_4A | NAIVE_4B
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/89 | 0/80 | 0/32 | 0/91 | 0/100 | 0/55 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/89 | 0/80 | 0/32 | 0/91 | 0/100 | 0/55 | 0/50
Other Adverse Events (participants affected / at risk) | 91/97 | 84/89 | 75/80 | 31/32 | 86/91 | 97/100 | 55/55 | 50/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 2H3H511_V (N=97) | 3H5_11_V (N=89) | 68_11_V (N=80) | 02_2_5_V (N=32) | 02_6_10_V (N=91) | NAIVE 123 (N=100) | NAIVE_4A (N=55) | NAIVE_4B (N=50)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/96 | 0 | 1/78 | 2 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0/96 | 0 | 0/78 | 0 | 27 | 0 | 1 | 20
Somnolence (Nervous system disorders) | 28/96 | 23 | 26/78 | 5 | 0 | 23 | 10 | 0
Chills (General disorders) | 0/96 | 0 | 0/78 | 0 | 23 | 0 | 0 | 7
Crying (General disorders) | 31/96 | 24 | 25/78 | 4 | 0 | 23 | 8 | 0
Injection site erythema (General disorders) | 61/96 | 63 | 42/78 | 22 | 57 | 65 | 38 | 37
Injection site induration (General disorders) | 48/96 | 48 | 33/78 | 15 | 44 | 48 | 28 | 25
Injection site pain (General disorders) | 84/96 | 80 | 71/78 | 31 | 84 | 94 | 55 | 48
Injection site swelling (General disorders) | 49/96 | 50 | 37/78 | 20 | 52 | 51 | 36 | 34
Malaise (General disorders) | 0/96 | 0 | 0/78 | 0 | 35 | 0 | 0 | 16
Pyrexia (General disorders) | 17/96 | 18 | 12/78 | 2 | 10 | 25 | 5 | 4
Eating disorder (Psychiatric disorders) | 31/96 | 32 | 30/78 | 5 | 0 | 36 | 13 | 0
Irritability (Psychiatric disorders) | 54/96 | 52 | 46/78 | 9 | 0 | 48 | 19 | 1
Diarrhoea (Gastrointestinal disorders) | 4/96 | 8 | 5/78 | 0 | 0 | 7 | 6 | 0
Nausea (Gastrointestinal disorders) | 0/96 | 0 | 0/78 | 0 | 12 | 0 | 0 | 8
Vomiting (Gastrointestinal disorders) | 5/96 | 6 | 2/78 | 1 | 0 | 10 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 13/96 | 1 | 3/78 | 5 | 10 | 8 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/96 | 0 | 0/78 | 0 | 18 | 0 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0/96 | 0 | 0/78 | 0 | 24 | 0 | 0 | 15
Pharyngitis (Infections and infestations) | 3/96 | 2 | 1/78 | 0 | 0 | 2 | 0 | 15
Tonsillitis (Infections and infestations) | 1/96 | 1 | 2/78 | 0 | 0 | 6 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.